CLINICAL TRIAL: NCT00051727
Title: Preventive Intervention for Mexican American Adolescents
Brief Title: Prevention of School Dropout for Mexican American Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R01MH064707 (NIH); R01MH064707 (NIH); DSIR 84-CTP
Record Dates: First submitted 2003-01-15; First posted 2003-01-17 (Estimated); Last update posted 2012-01-10 (Estimated); Status verified 2012-01

CONDITIONS: Depression; Conduct Disorder
MeSH Terms: conditions — Depression; Conduct Disorder

INTERVENTIONS:
Behavioral: Bridges to High School Project

SUMMARY:
The purpose of this study is to test the efficacy of a family-based psychosocial intervention to prevent school disengagement and reduce the incidence of depression, conduct disorders, and school dropout for Mexican American adolescents.

DETAILED DESCRIPTION:
Mexican American adolescents are at an increased risk for interrelated problems of poor mental health and school dropout. Unfortunately, there is a lack of interventions specifically designed to address this risk. This study will evaluate a preventive intervention for low-income Mexican American adolescents.

Participants are randomly assigned to either a multi-component intervention called the Bridges to High School Program or a Low Dose Workshop. The 11-week multi-component intervention takes place during the fall semester of seventh grade and consists of an adolescent group, a parenting group, a combined (parent-adolescent) family group, and a school liaison. This intervention focuses on adolescent coping skills, parenting practices, family cohesion, and parental support for education. The Low-Dose Workshop consists of a 3-hour workshop in which adolescents and parents are given information and resources to facilitate school engagement. Participants are assessed prior to and immediately following the intervention and again in eighth and ninth grade. Academic and mental health outcomes are measured with questionnaire-based interviews given to caregivers and adolescents. Teachers are asked to complete questionnaires; archival school data are also collected. Diagnostic interviews are conducted at the ninth grade assessment.

ELIGIBILITY:
Inclusion criteria:

* Mexican American adolescent with at least one primary caregiver
* Enrolled in seventh grade in one of four inner-city schools
* Adolescent and participating caregivers must be able to receive intervention in the same language (English or Spanish)

Exclusion criteria:

* High risk for suicide

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 480
Dates: Start 2002-10

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Gonzales, Ph.D., Principal Investigator — Arizona State University
Locations (1):
- Prevention Research Center, Arizona State University, Tempe, Arizona, United States